CLINICAL TRIAL: NCT04347642
Title: Umbilical vs Paraumbilical Trocar Placement in Patients Undergoing Elective Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Clinical Professor, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Garcilaso 2020/1
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical port (Active Comparator): A Hasson port will be inserted at the level of the umbilicus,in the midline, traversing only aponeurotic layers.
  Interventions: Procedure: Umbilical port placement
- Paraumbilical port (Experimental): A bladeless 12mm port will be inserted lateral to the midline, traversing aponeurotic layers and rectus abdominis muscle.
  Interventions: Procedure: Paraumbilical port placement

INTERVENTIONS:
Procedure: Umbilical port placement — The port will be inserted in the midline at the level of the umbilicus.
  Arms: Umbilical port
Procedure: Paraumbilical port placement — The port will be inserted 3-4cm laterally to the midline at the level of the umbilicus.
  Arms: Paraumbilical port

SUMMARY:
The aim of this study will be to assess the incisional hernia rate of umbilical or paraumbilical port 12 months after laparoscopic cholecystectomy.

Patients will be randomized into 2 groups:

* G1: 12mm Umbilical port will be inserted in the umbilical region, with open access and using a Hasson port
* G2: 12 mm paraumbilical port will be inserted laterally to the midline, with close access and using and optical port.

Incisional hernia at the level of this port insertion will be assessed by physical examination and, in case of doubst, by ultrasonography, 12 months after surgery.

DETAILED DESCRIPTION:
The aim of this study will be to assess the incisional hernia rate of umbilical or paraumbilical port 12 months after laparoscopic cholecystectomy.

Patients will be randomized into 2 groups:

* G1: 12mm Umbilical port will be inserted in the umbilical region, with open access and using a Hasson port. Pneumoperitoneum will be done by this Hasson port.
* G2: 12 mm paraumbilical port will be inserted laterally to the midline, with close access and using and optical port, traversing the rectus abdominal muscle. Pneumoperitoneum will be previously done using a Veress needle.

Incisional hernia at the level of this port insertion will be assessed by physical examination and, in case of doubst, by ultrasonography, 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic cholecystectomy
* Acceptance to participate in the study and sign of informed consent form

Exclusion Criteria:

* A gallstone larger than 10mm observed at preoperative ultrasonography
* Coexistence of umbilical hernia or previous umbilical hernioplasty
* Previous laparotomy involving the umbilical region
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia at the level of the trocar insertion | 12 months after surgery
  The incisional hernia at the level of the umbilical or paraumbilial trocar insertion will be assessed by physical examination, or with ultrasonography in case of doubts.

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto Gonzalez, Study Chair — Centro PDH
Locations (2):
- Gilberto Gonzalez, Guadalajara, Mexico
- Jaime Ruiz-Tovar, Madrid, Introducir Provincia O Estado, Spain

IPD SHARING:
Plan to Share IPD: No